CLINICAL TRIAL: NCT07119424
Title: Multidisciplinary Dissection of Renal and Metabolic Effects of Glyfozines on Elderly Patients: From Molecular Aspects to Clinical Indications
Status: Recruiting | Type: Observational
Sponsor: Chiara Lanzani (Other)
Responsible Party: Sponsor-Investigator, Chiara Lanzani, Professor, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: PNRR-MCNT2-2023-12377474
Record Dates: First submitted 2025-07-01; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Elderly Patients (>65 Years); Diabetes (DM); Heart Disease; Renal Diseases; Internal Disease
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Kidney Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with Nephrological, Diabetologic, Cardiological and Internal diseases: Patients aged ≥65 years, either females or males, who have just been prescribed, in accordance with clinical practice and due to clinical reasons independent of the study, a SGLT2i for any clinical indication for SGLT2i use, who have not yet started SGLT2i therapy, and yet not under SGLT2i treatment.

SUMMARY:
The project aims to study the impact of SGLT2i therapy on clinical and biochemical aspects. in elderly. The project will combine different types of data, such as clinical and biological information, and will use advanced Bayesian statistical methods to understand the relationship between risk factors and patient outcomes following treatment with SGLT2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study;
2. Patients must be enrolled also in MED-Cli e MED-Mol studies by signing both the MED-Cli e MED-Mol informed consents.
3. The medical product is the standard of care for the patient and has been prescribed according to clinical practice and independent of the present study;
4. Age ≥65 years;
5. Participant has not yet started the prescribed SGLT2i therapy;
6. Participant has at least one clinical indication for SGLT2i use according to clinical practice guidelines.

Exclusion Criteria:

1. Current or previous use of SGLT2i;
2. Inability to sign the informed consent.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged ≥65 years, either females or males, who have just been prescribed, in accordance with clinical practice and due to clinical reasons independent of the study, a SGLT2i for any clinical indication for SGLT2i use, who have not yet started SGLT2i therapy, and yet not under SGLT2i treatment. Patients must be enrolled also in MED-Cli e MED-Mol studies by signing both the MED-Cli e MED-Mol informed consents.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Patient health status prior and after 6 months of SGLT2i therapy through Frailty Index variation (FI) | From enrollment to 6 months
  Patient health status prior and after 6 months of SGLT2i therapy through Frailty Index variation (FI).
  The FI is score measured by comparing the ratio of health deficits present within an individual to possible health deficits, using a pre-specified list of 30 or more deficits.
  Deficits included in the model will be collected during the visit trough questionnaires and clinical and biochemical evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided